CLINICAL TRIAL: NCT02858427
Title: Cognitive Inhibition Impairment and Suicide Attempt in Elderly: Eye Tracking Characterization and Impact of Psychosocial Interactions
Brief Title: Cognitive Inhibition, Psychosocial Interactions and Suicide Attempt in Elderly
Acronym: OBSUIVAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: P/2016/288
Record Dates: First submitted 2016-08-01; First posted 2016-08-08 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Suicide
Keywords: cognitive inhibition; elderly; suicide attempt; depression
MeSH Terms: conditions — Suicide; Suicide, Attempted; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- depressed with suicide attempt (SA) (Experimental): elderly depressed patients with a history of suicide attempt. interventions: eye tracking, neuropsychological assessment, psychiatric assessment and sociological interview.
  Interventions: Behavioral: eye tracking; Behavioral: neuropsychological assessement; Behavioral: psychiatric assessment; Behavioral: sociological interview
- depressed without a history of SA (Experimental): elderly depressed patients without a history of suicide attempt. interventions: eye tracking, neuropsychological assessment, psychiatric assessment and sociological interview.
  Interventions: Behavioral: eye tracking; Behavioral: neuropsychological assessement; Behavioral: psychiatric assessment; Behavioral: sociological interview

INTERVENTIONS:
Behavioral: eye tracking — several oculomotor parameters will be recorded using vide-oculography techniques (eye tracking) trough different tasks: saccade, antisaccade, and picture scanning.
  Saccade task: the patient is looking at a screen and is asked to fix his gaze as quickly and accurately as possible on the red dot appearing on the periphery of the screen.
  Prosaccade task: the patient is looking at a screen and is asked to fix his gaze as quickly and accurately as possible on the opposite side relative to the red dot appearing on the periphery of the screen.
  Picture Scanning: participant is instructed to freely watch pictures with different emotional valence.
Behavioral: neuropsychological assessement — the neuropsychological assessment aims to identify any impairment of executive functioning through several tasks: Mini mental state examination (mmse), isaac set test (STI) trail making test (TMT A and B), Grober test, Stroop test, verbal fluency, Go No Go task, memory impairment screen (MIS), picture naming test (DO30), copying figure test, digit span and categorical matching test.
Behavioral: psychiatric assessment — this evaluation aims to characterize the mental status of the patient. Different scales will be used: Montgomery and ASberg depression rating scale (MADRS), Columbia-suicide severity rating scale (C-SSRS), Beck depression inventory (BDI), Barratt impulsiveness scale (BIS-10), Buss and Durkee Hostility Inventory (BDHI), Balloon, analogue risk task (BART), Iowa gambling task (IGT), and Childhood trauma questionnaire (CTQ).
Behavioral: sociological interview — this interview aims to characterize social interactions of the patients, their duration, their evolution and the perception of each participant on this subject.

SUMMARY:
The study aims to determine the correlation between the cognitive inhibition impairment and the history of suicide attempt in elderly depressed patients.

DETAILED DESCRIPTION:
2 groups of patients will be studied: in the first group, depressed patients with a history of suicide attempt will be included whereas in the second group, depressed patients without a history of suicide attempt will be included.

For each group, the cognitive inhibition will be assessed trough an eye tracker task (antisaccade).

Both groups will also be compared on their neuropsychological characteristics and the quality of social interactions of participants.

ELIGIBILITY:
Inclusion Criteria:

* major depressive disorder according to Diagnostic ans Statistical Manual (DSM) V
* group 1: with a history of suicide attempt
* group 2: without a history of suicide attempt

Exclusion Criteria:

* other psychiatric disease
* guardianship

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-02-06 (Actual); Primary Completion 2019-08-06 (Estimated); Study Completion 2020-02-06 (Estimated)

PRIMARY OUTCOMES:
antisaccade error rate | 1 month max. after inclusion

SECONDARY OUTCOMES:
saccade accuracy | 1 month max. after inclusion
  distance between the eye position at the end of the first saccade, and the ideal position to engage the target in central vision
saccadic intrusion | 1 month max. after inclusion
  gaze deviation into a saccade greater than 3° during visual fixation
maximal speed of the gaze | 1 month max. after inclusion
  maximum speed of visual tracking without triggering any saccade
saccade reaction time | 1 month max. after inclusion
fixation duration on pictures | 1 month max. after inclusion
social interaction quality score | 6 month max. after inclusion

OTHER OUTCOMES:
neuropsychological test score | 1 month max. after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: pierre vandel, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (2):
- France (2):
  - CHU Besancon, Besançon, Doubs
  - CHS Bavilliers, Bavilliers

IPD SHARING:
Plan to Share IPD: No